CLINICAL TRIAL: NCT01927744
Title: Randomized, Placebo-Controlled, Phase 2 Study Of Induction Chemotherapy With Cisplatin/Carboplatin, And Docetaxel With Or Without Erlotinib In Patients With Head And Neck Squamous Cell Carcinomas Amenable For Surgical Resection
Brief Title: Study of Chemotherapy With Cisplatin/Carboplatin, and Docetaxel With or Without Erlotinib in Patients With Head and Neck Squamous Cell Carcinomas Amenable for Surgical Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Astellas Pharma Inc (Industry); The Kadoorie Charitable Foundations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0179; NCI-2014-01390 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Squamous cell carcinoma of the head and neck; SCCHN; Oral cavity squamous cell carcinomas; Docetaxel; Taxotere; Erlotinib; Erlotinib Hydrochloride; OSI-774; CP358774; Tarceva; Questionnaire; Survey; Phone call
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Erlotinib Hydrochloride; Surveys and Questionnaires; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chemotherapy + Erlotinib (Experimental): Docetaxel 75 mg/m2 by vein followed by Cisplatin 75 mg/m2 or Carboplatin AUC 6 mg.min/ml by vein on Day 1 of each 21 day cycle for a maximum of 3 cycles, plus Erlotinib 150 mg by mouth daily continuously until the day before surgery. Questionnaire completion at baseline, 14 days after treatment completion, and 8 weeks after surgery. Phone call made to patient 1 time each year after the end of treatment visit.
  Interventions: Drug: Docetaxel; Drug: Erlotinib; Behavioral: Questionnaires; Behavioral: Phone Call; Drug: Chemotherapy
- Chemotherapy + Placebo (Experimental): Docetaxel 75 mg/m2 by vein followed by Cisplatin 75 mg/m2 or Carboplatin AUC 6 mg.min/ml by vein on Day 1 of each 21 day cycle for a maximum of 3 cycles, plus placebo 150 mg by mouth daily continuously until the day before surgery. Questionnaire completion at baseline, 14 days after treatment completion, and 8 weeks after surgery. Phone call made to patient 1 time each year after the end of treatment visit.
  Interventions: Drug: Docetaxel; Other: Placebo; Behavioral: Questionnaires; Behavioral: Phone Call; Drug: Chemotherapy

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 by vein on Day 1 of each 21 day cycle for a maximum of 3 cycles.
  Other Names: Taxotere
Drug: Erlotinib — 150 mg by mouth daily continuously until the day before surgery.
  Other Names: Erlotinib Hydrochloride; OSI-774; CP358774; Tarceva
  Arms: Chemotherapy + Erlotinib
Other: Placebo — 150 mg by mouth daily continuously until the day before surgery.
  Arms: Chemotherapy + Placebo
Behavioral: Questionnaires — Questionnaire completion at baseline, 14 days after treatment completion, and 8 weeks after surgery.
  Other Names: Surveys
Behavioral: Phone Call — Phone call made to patient 1 time each year after the end of treatment visit.
Drug: Chemotherapy — Cisplatin 75 mg/m2 or Carboplatin AUC 6 mg.min/ml by vein on Day 1 of each 21 day cycle for a maximum of 3 cycles.

SUMMARY:
The goal of this clinical research study is to learn if adding erlotinib to a standard chemotherapy combination (docetaxel and either cisplatin or carboplatin) can help to control SCCHN. The safety of this drug combination will also be studied.

In this study, erlotinib will be compared to a placebo. A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

This is an investigational study. Erlotinib is approved by the FDA for treatment of non-small cell lung cancer. Its use in this study is experimental. Docetaxel, cisplatin, and carboplatin are all FDA approved and commercially available for the treatment of SCCHN.

Up to 100 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups (also known as an Arm):

* If you are in Arm A, you will receive standard chemotherapy in combination with erlotinib.
* If you are in Arm B, you will receive standard chemotherapy in combination with a placebo.

If you are 1 of the first 30 patients to be enrolled on the study, you will have an equal chance of being assigned to either group. If you are one of the next 20 patients to be enrolled on the study, you will have a higher chance of being assigned to the group that appears to be performing better. Up to 50 more participants will then be assigned to a study group based on the results seen in the first 50 participants.

Neither you nor the study doctor will know if you are receiving erlotinib or placebo. However, if needed for your safety, the study doctor will be able to find out what you are receiving.

Study Drug Administration:

You will receive docetaxel and either cisplatin or carboplatin by vein on Day 1 of up to 3 study cycles, over about 1-2 hours. The study doctor will tell you whether you are receiving cisplatin or carboplatin. Each study cycle will be 3 weeks.

You will also take tablets of either erlotinib or placebo every day until (and including) the day before your scheduled surgery. You should take the tablets with about 1 cup (8 ounces) of water. You should take the tablet on an empty stomach, at least 1 hour before or 2 hours after a meal. You should take the tablet at around the same time each day, preferably in the morning. Your eating habits around the time you take the tablet should stay the same while you are on study. lf you vomit, and you can actually see the tablet, you may take another tablet. If not, you should not take another tablet until your next scheduled dose.

You will continue to take erlotinib or placebo daily until the day prior to surgery (including the day prior to surgery).

You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Visits:

On Day 1 of each Cycle, you will receive the study drugs, as described above.

Within 7 days before Cycles 2 and 3:

* You will have a physical exam.
* You will be asked about your current smoking status and tobacco use.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

At least 14 days after the last dose of chemotherapy:

* You will have a physical exam.
* You will be asked about your current smoking status and tobacco use.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* You will have an MRI or CT scan of the head and neck. If the study doctor thinks it is needed, additional imaging scans may be performed.
* You will complete a questionnaire about how you feel about different aspects of your daily life. It should take you about 15 minutes to complete the questionnaire.
* Blood (about 1-2 teaspoons) will be drawn for biomarker and pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points.

At any point while you are on study, if you can become pregnant and your doctor thinks it is needed, you will have a blood (about 1 teaspoon) or urine pregnancy test.

Surgery:

After you stop taking the study drug/placebo, you will have the surgery you were already scheduled to receive. You will sign a separate consent form that describes the surgery and its risks. As part of this study, tumor tissue will be collected during the surgery and checked for the status of the disease as well as any spread of the disease.

Length of Study:

You may receive the standard chemotherapy combination for up to 3 cycles. You may take the study drug/placebo up until the day before surgery. If you have side effects from the chemotherapy, it is possible that you may stop taking the chemotherapy combination and continue to receive the study drug/placebo up until surgery. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your active participation on the study will be over after the end-of-treatment visit.

End of Treatment Visit:

About 8 weeks after surgery, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 1-2 teaspoons) will be drawn for biomarker and PK testing.
* You will complete the questionnaire about your daily life.
* If you can become pregnant and your doctor thinks it is needed, you will have a blood (about 1 teaspoon) or urine pregnancy test.

Long Term Follow Up:

After the end of treatment visit, you will be called at least 1 time each year to check on how you are doing. You (or your family members or designees) may be contacted by telephone, in writing, by e-mail, or during clinic visits. It is important to keep your contact information up to date with the study staff. This information may also be collected by checking your medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or histologically/citologically confirmed HNSCC of the oral cavity, stage III, IVA or IVB (according to the AJCC 7th edition). Patients with a suspected lesion may be enrolled and a baseline biopsy will be obtained as part of the study. If squamous cell histology is not confirmed, patients will be discontinued from the study.
2. Patients must have surgically resectable disease, in the opinion of the treating physician
3. Age ≥ 18 years.
4. ECOG PS ≤ 2 (Appendix C)
5. Adequate bone marrow, hepatic and renal function defined by: 6. ANC ≥ 1.5 x 109/L;

7. Platelet count ≥ 100 x 109/L;

8. ALT (SGPT) ≤ 1.5 x upper limit of normal (ULN);

9. Total bilirubin ≤ ULN (patient's with Gilbert's syndrome are eligible, even if total bilirubin is > ULN);

10. Alkaline phosphatase ≤ 2.5 x ULN;

11. Serum creatinine ≤ 1.5 x ULN.

12. Patients with reproductive potential (e.g., females menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures for the duration of study drug therapy and for at least 30 days after completion of study drug therapy. Female patients of childbearing potential must provide a negative pregnancy test (serum or urine) ≤ 14 days prior to treatment initiation.

13. Written informed consent to participate in the study according to the investigational review board (IRB).

Exclusion criteria:

1. Histology other than squamous cell carcinoma.
2. Primary sites other than oral cavity.
3. Prior chemotherapy or biologic therapy for the same HNSCC. Prior chemotherapy or biologic therapy for a different previous HNSCC is allowed
4. History of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g., Crohn's disease, ulcerative colitis). Patients requiring feeding tubes are permitted
5. Other active solid malignancies within 2 years prior to randomization, except for basal cell or squamous cell skin cancer or in situ cervical or breast cancer or superficial melanoma.
6. Serious underlying medical condition which would impair the ability of the patient to receive protocol treatment, in the opinion of the treating physician.
7. History of allergic reactions to compounds of similar chemical composition to the study drugs (docetaxel, cisplatin, carboplatin, erlotinib or their excipients), or other drugs formulated with polysorbate 80.
8. Any concurrent anticancer therapy, excluding hormonal therapy for prostate or breast cancer.
9. Women who are pregnant or breast-feeding and women or men not practicing effective birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiuning Le, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with suspected or histologically/citologically confirmed HNSCC of the oral cavity, stage III, IVA or IVB (according to the AJCC 7th edition) are enrolled. Patients with a suspected lesion may be enrolled and a baseline biopsy will be obtained as part of the study. Must be age ≥ 18 years. ECOG PS ≤ 2 (Appendix C) and adequate bone marrow, hepatic and renal function defined by: 6. ANC ≥ 1.5 x 109/L.
Pre-assignment Details: A total of 55 participants were enrolled. Three participants did not proceed to randomization: two were screen failures and one was lost to follow-up prior to treatment initiation. The remaining 52 participants were randomized.
Period: Overall Study
Arm/Group | Chemotherapy + Erlotinib | Chemotherapy + Placebo
Started | 24 | 28
Completed | 22 | 19
Not Completed | 2 | 9
Not completed — Death | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy + Erlotinib | Chemotherapy + Placebo | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Continuous [Median (Full Range); unit: years] | 60 [29 to 74] | 57 [26 to 71] | 58 [26 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 14 | 17 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 22 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 24 | 28 | 52

OUTCOME MEASURES:

1. Primary Outcome: Major Pathologic Response (MPR) Rate (Primary (Overall) Analysis)
Description: Major Pathologic Response (MPR) was defined as ≤ 10% residual biable tumor cells in the resected primary tumor specimen following completion of neadjuvant therapy.
Time Frame: At surgery following completion of induction chemotherapy (up to approximately 63 days after treatment initiation).
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Erlotinib | Chemotherapy + Placebo
Number analyzed (Participants) | 23 | 24
participants | 7 | 10

ADVERSE EVENTS:
Time Frame: Up to 9 weeks (from initiation of induction chemotherapy through surgery).
Description: MedDRA v12
Arm/Group | Chemotherapy + Erlotinib | Chemotherapy + Placebo
All-Cause Mortality (participants affected / at risk) | 2/24 | 9/28
Serious Adverse Events (participants affected / at risk) | 8/24 | 10/28
Other Adverse Events (participants affected / at risk) | 23/24 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Erlotinib (N=24) | Chemotherapy + Placebo (N=28)
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0
Cardiac (Cardiac disorders) | 0 | 0
Cytopenia (Blood and lymphatic system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 0 | 0
Fatigue (General disorders) | 0 | 5
Gastroninstenal Disorders (Gastrointestinal disorders) | 3 | 2
Hearing (Ear and labyrinth disorders) | 0 | 0
Infection (Infections and infestations) | 2 | 1
Metabolic and Nutrition (Metabolism and nutrition disorders) | 6 | 1
Nausea and Vomiting (Gastrointestinal disorders) | 5 | 2
Other (General disorders) | 1 | 2
Pain (General disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0
Any AE (General disorders) | 8 | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Erlotinib (N=24) | Chemotherapy + Placebo (N=28)
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 15
Cardiac (Cardiac disorders) | 4 | 1
Cytopenia (Blood and lymphatic system disorders) | 9 | 5
Dizziness (Nervous system disorders) | 11 | 6
Fatigue (General disorders) | 19 | 16
Gastroninstenal Disorders (Gastrointestinal disorders) | 16 | 20
Hearing (Ear and labyrinth disorders) | 0 | 3
Infection (Infections and infestations) | 10 | 4
Metabolic and Nutrition (Metabolism and nutrition disorders) | 9 | 8
Nausea and Vomiting (Gastrointestinal disorders) | 16 | 15
Other (General disorders) | 16 | 14
Pain (General disorders) | 8 | 15
Rash (Skin and subcutaneous tissue disorders) | 19 | 14
Any AE (General disorders) | 23 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT01927744/Prot_SAP_001.pdf
  • Informed Consent Form (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT01927744/ICF_000.pdf